CLINICAL TRIAL: NCT03194438
Title: Feasibility and Acceptability of an Integrative Therapy for Symptom Management in Persons With Pulmonary Hypertension
Brief Title: Urban Zen Integrative Therapy for Persons With Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017H0022
Record Dates: First submitted 2017-06-15; First posted 2017-06-21 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Hypertension; Chronic Disease
Keywords: Pulmonary Hypertension; Symptom Management; Behavioral Intervention; Integrative Therapy; Quality of Life
MeSH Terms: conditions — Hypertension, Pulmonary; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Single cohort of sample with repeated measure assessment of symptoms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UZIT arm (Experimental): Multi-modal components integrative therapy intervention program, Urban Zen Integrative Therapy.
  Interventions: Behavioral: Urban Zen Integrative Therapy (UZIT)

INTERVENTIONS:
Behavioral: Urban Zen Integrative Therapy (UZIT) — Multi-modal components integrative therapy program (UZIT) that includes essential oil, gentle body movement, body-awareness meditation, and Reiki.

SUMMARY:
The primary goal of this study is to determine the feasibility and acceptability of a 6-week multicomponent integrative therapy program, Urban Zen Integrative Therapy (UZIT), for adults with chronic, life-limiting cardiopulmonary disease. The secondary goal is to determine preliminary efficacy of UZIT in symptom management. Pulmonary hypertension (PH) presents an excellent model of a severe, life-limiting cardiopulmonary condition with high symptom burden and poor outcomes suitable for this scientific inquiry. Despite medical and pharmacological advances in the treatment, 50-55% of persons with PH will die within three years after diagnosis. Medical management often involves life-long complex pharmacological treatment requiring high levels of skill, knowledge, and social support. Clusters of bothersome symptoms such as chest pain, anxiety, insomnia, dyspnea, and fatigue can overwhelm patients' ability to manage daily activities and medication treatment regimens. Side effects of treatment induce additional noxious symptoms. The high prevalence of physical symptoms, depression, and anxiety among adults with PH confirmed in our prior work, can also lead to reduced (HRQoL). A literature search found no published report of complementary, integrative therapy interventions to alleviate symptoms in adults with PH. This study will use a single group repeated-measures design to address the feasibility and acceptability of the intervention and to explore preliminary efficacy.

DETAILED DESCRIPTION:
This feasibility and acceptability study will use a pre/post intervention (6-weeks UZIT program) mixed-method design with repeated (weekly) measures of a single cohort of 20 patients with PH. This study will also explore preliminary efficacy testing to construct sample size estimates for future randomized control trials. Patients will serve as their controls.

This study will enroll 20 patients from two PH clinics within the Ohio State University Wexner Medical Center (OSUWMC). Patients with PH condition related to the cardiac cause are managed at the OSU Cardiology clinic located at the Ross Heart Hospital. Patients with PH condition related to other causes are managed at the OSU Pulmonary clinic at Martha Morehouse. These inter-professional clinics provide access to a patient population with diverse race/ ethnicity, sex, and age. All eligible patients managed at both PH clinics at OSUWMC will be invited to participate. Patients in both clinics receive standard medical treatments according to institutional and national clinical practice guidelines.

ELIGIBILITY:
Inclusion criteria are:

1. confirmed diagnosis of PH in the past 1 year,
2. age > 18 years, (children typically have different etiologies, and often require parent involvement in symptom management),
3. ability to ambulate independently,
4. New York Heart Association functional classification II/III, and
5. willingness to participate in the entire 6-8 weeks study.

Exclusion criteria are

1. known allergies to essential oils (lavender, lemon, or peppermint),
2. Asthma condition,
3. psychiatric illness requiring hospitalization within the last year per self-report or medical record,
4. self-reported pregnancy,
5. on-going participation in mind-body integrative therapy, and
6. inability to read/write English (to complete questionnaires).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tania VonVisger, PhD, Principal Investigator — SUNY Buffalo
Locations (1):
- The Ohio State University Ross Heart Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Von Visger TT, Thrane SE, Klatt MD, Chang YP, Happ M. Deep Relaxation Experience with Complementary Urban Zen Integrative Therapy: Qualitative Thematic Analysis. West J Nurs Res. 2021 Aug;43(8):723-731. doi: 10.1177/0193945920973941. Epub 2020 Nov 27. PMID 33246388
- [Derived] Von Visger TT, Thrane SE, Klatt MD, Dabbs AD, Chlan LL, Tan A, Happ MB. The Impact of Urban Zen Integrative Therapy on Symptoms and Health-Related Quality of Life for Patients with Pulmonary Hypertension. J Palliat Med. 2020 May;23(5):703-711. doi: 10.1089/jpm.2019.0359. Epub 2019 Oct 31. PMID 31644380

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UZIT Arm
Started | 14
Completed | 12
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | UZIT Arm
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.26 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White | 11
  Black | 3
  Non-Hispanic or Latino | 13
  Latino | 1
Region of Enrollment [Number; unit: participants]
  United States | 14
Pulmonary Arterial Hypertension Symptom Scale - SOB Exertion [Mean (Standard Deviation); unit: units on a scale] — Measures pulmonary hypertension-related symptom severity. Minimum score 0, maximum score 10, with 10 being the worst outcome. There are no sub-scores in this measure.
  units on a scale | 6.70 (2.26)
Cambridge Pulmonary Hypertension Outcome Review - Symptom Burden [Mean (Standard Deviation); unit: units on a scale] — Measures pulmonary hypertension-related Quality of Life: Sub- scales -
  Symptom Severity Scale Minimum score 0, maximum score 25, with 25 being the worst outcome.
  units on a scale | 12.00 (5.24)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Arterial Hypertension Symptom Scale - SOB With Exertion
Description: Symptoms assessment and Health-related quality of life assessment. We focused on the shortness of breath. The minimum and maximum scores are 0 and 10, respectively. A higher score indicates the worst outcome.Measured at baseline and 6-weeks post-intervention for comparision
Time Frame: Baseline and 6-week post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UZIT Arm
Number analyzed (Participants) | 9
units on a scale | 3.0 (2.54)

2. Secondary Outcome: Change in Cambridge Pulmonary Hypertension Outcome Review.
Description: This instrument was used to measure the overall Health-related quality of life with multiple domains. We focused on the Symptom Burden domain.
  The minimum and maximum scores range from "0" to "25", indicating "good" and "poor" symptom burden, respectively.
  The scale of the change score indicates the level of MID (minimum importance difference). If the score is more significant than 2.0 MID, the intervention makes a minimal level of importance in their quality of life perception.
  Measurements were taken at baseline and 6-weeks post-intervention for comparision.
Time Frame: Baseline and 6-week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UZIT Arm
Number analyzed (Participants) | 9
score on a scale | 8.91 (5.24)

ADVERSE EVENTS:
Time Frame: Each participant spent 6 weeks in the study, adverse event data were collected over that 6 week period.
Description: The definition of adverse event and/or serious adverse event used did not differ from the clinicaltrials.gov definitions.
Arm/Group | UZIT Arm
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
The final analysis for PAHSS and CAMPHOR were obtained from 9 participants who completed the entire 6-week intervention and with complete assessment data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT03194438/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT03194438/ICF_001.pdf